CLINICAL TRIAL: NCT00735293
Title: The Use of the VASER System in the Treatment of Axillary Hyperhidrosis and/or Axillary Bromidrosis
Brief Title: VASER Treatment of Axillary Hyperhidrosis/Bromidrosis
Acronym: VASER AxHH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Commons Aesthetic Plastic Surgery (Other)
Collaborators: Sound Surgical Technologies, LLC. (Industry)
Responsible Party: George W. Commons, M.D., Commons Aesthetic Plastic Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VASER AxHH
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Axillary Hyperhidrosis
Keywords: hyperhidrosis; bromidrosis; bromhidrosis; osmidrosis; hircismus; excessive; underarm; sweat; perspiration; Body Odor
MeSH Terms: conditions — Hyperhidrosis; Body Odor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): There is only one arm to this study. All patients will receive treatment with the VASER for their axillary hyperhidrosis/bromidrosis
  Interventions: Device: VASER

INTERVENTIONS:
Device: VASER — A small incision will be made in the underarm. A VASER probe will be inserted under the skin to break apart fat and sweat glands under the skin. A small hollow tube will be used to draw out the broken-down skin and the incision will be closed with a stitch.
  Other Names: Sound VASER System

SUMMARY:
Patients with excessive underarm odor and sweating and/or odor are treated with the VASER system to determine the VASER's effectiveness in reducing underarm sweat and odor

DETAILED DESCRIPTION:
Patients with excessive underarm sweat and/or odor are recruited. The effect that excessive underarm sweat and/or odor has on their lifestyle is evaluated. They are surgically treated with the VASER system and followed up for 6 months to evaluate side effects, adverse events and effectiveness. Additional lifestyle evaluations are completed for comparison to pre-surgery answers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to appear for all scheduled, post-operative visits
* Have axillary hyperhidrosis/bromidrosis that does not respond to conventional, non-invasive treatment

Exclusion Criteria:

* under the age of 18
* have undergone a prior surgical intervention for treatment of axillary hyperhidrosis (e.g.) Skoog procedure, ETS)
* have been treated with a systemic or topical agent for axillary hyperhidrosis in the past 30 days
* are deemed inappropriate candidates for surgery due to medical or mental health reasons
* are currently being treated with investigational agents or have participated in an investigational study within 60 days prior to surgery
* elect not to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of the VASER for treatment of axillary hyperhidrosis using patient self-report assessments | 6 months
To assess the effectiveness of the VASER for the treatment of axillary bromidrosis using patient self report assessment | 6 months

SECONDARY OUTCOMES:
To assess patient's post-operative pain level following VASER using patient self report assessments. | 2 months
To assess patients healing time following VASER treatment of axillary hyperhidrosis | 6 months
To establish safe and effective procedural guidelines and surgical endpoints for the treatment of axillary hyperhidrosis using the VASER | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Commons Aesthetic Plastic Surgery, Palo Alto, California, United States

REFERENCES:
- See also: Sound VASER System — http://vaser.com